CLINICAL TRIAL: NCT06671743
Title: Effect of Premedication on Post-endodontic Pain in Patients With Symptomatic Irreversible Pulpitis, a Triple-blinded Randomized Control Trial
Brief Title: Premedication on Post-endodontic Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-COD-STD-22-JULY-2024
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Premedication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- trypsin-chymotrypsin (Experimental)
  Interventions: Procedure: Root canal treatment
- Ibuprofen (Active Comparator)
  Interventions: Procedure: Root canal treatment
- paracetamol (Active Comparator)
  Interventions: Procedure: Root canal treatment
- placebo (Placebo Comparator)
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Root canal treatment — History of presenting illness will be recorded and vitality testing will be done in addition to pre-operative radiograph.
  Patient will read and sign the consent form. Pre-operative pain score will be recorded using visual analogue scale. The patient will take the preoperative medication 1 hour prior to the procedure.
  The patient will receive 1 cartridge of LA with inferior alveolar nerve block (2% lidocaine 1:80000) and a rubber dam will be used for isolation.
  Access cavity will be prepared and working length will be determined. Cleaning and shaping of the root canal system will be performed followed by obturation using a standardized protocol followed by final coronal restoration.
  Postoperative pain score will be recorded at the 6, 12, 24, and 48 hours using visual analogue pain scale.

SUMMARY:
The goal of this clinical trial is to compare the efficacy of preoperative administration of alpha-chemo-trypsin, ibuprofen, and acetaminophen in managing post-endodontic pain in patients with symptomatic irreversible pulpitis. The main question it aims to answer is:

What is the efficacy of preoperative administration of alpha-chemo-trypsin, ibuprofen, and acetaminophen in managing post-endodontic pain in patients with symptomatic irreversible pulpitis? Participants will undergo root canal treatment after premedication. Researchers will compare [alpha-chemo-trypsin, ibuprofen, and acetaminophen] to see the intensity of post-endodontic pain.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for root canal treatment Patients diagnosed with symptomatic irreversible pulpitis with normal apical tissue in mandibular molars

Exclusion Criteria:

* • Patient under any medication or analgesic intake for pain management.

  * Patients with any systemic health issues
  * Patient allergies to trypsin-chymotrypsin, ibuprofen, and paracetamol
  * Pregnancy.
  * Non-restorable teeth.
  * Immature roots.
  * Calcifications.
  * Resorptions.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Post-endodontic pain score | 6 hours
  Post operative pain score will be recorded using the visual analogue pain scale, where the patient will mark a point on a 10-cm line representing a continuum from 'no pain' to 'worst pain imaginable.
Post-endodontic pain score | 12 hours
  Post operative pain score will be recorded using the visual analogue pain scale, where the patient will mark a point on a 10-cm line representing a continuum from 'no pain' to 'worst pain imaginable.
Post-endodontic pain score | 24 hours
  Post operative pain score will be recorded using the visual analogue pain scale, where the patient will mark a point on a 10-cm line representing a continuum from 'no pain' to 'worst pain imaginable.
Post-endodontic pain score | 48 hours
  Post operative pain score will be recorded using the visual analogue pain scale, where the patient will mark a point on a 10-cm line representing a continuum from 'no pain' to 'worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided